CLINICAL TRIAL: NCT05284916
Title: Difference in Patterns of Liver Diseases Related Admissions in Sohag University Hospital After the Era of Direct Acting Antiviral Drugs
Brief Title: Difference in Patterns of Liver Diseases Related Admissions After the Era of DAAS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Momena Hassan Ahmed, Tropical medicine and gastroenterology department, Sohag University
Other Study IDs: Soh-Med-22-03-09
Record Dates: First submitted 2022-03-10; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Patternsof Liver Diseasesadmissions After Era of DAAS

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients admitted at Sohag University Hospital diagnosed with liver diseases: The study will be conducted in two stages. The first one is a retrospective collection of the data from patients records during the period from Feburary 2017 to January 2018 and the second stage will include agroup of patients that will be admitted to Tropical Medicine and Gastroenterology Department within 6months after protocol acceptance
  Interventions: Behavioral: liver diseases admissions

INTERVENTIONS:
Behavioral: liver diseases admissions — The different patterns of liver disease related admissions after the era of DAAS

SUMMARY:
Liver disease accounts for approximately 2 million deaths per year worldwide, 1 million due to complications of cirrhosis and 1 million due to viral hepatitis and hepatocellular carcinoma Hepatitis is defined as inflammation of the liver that can result from a variety of causes such as heavy alcohol use, autoimmune, drugs, or toxins In the United States, the most common types of viral hepatitis are Hepatitis A, Hepatitis B, and Hepatitis C The other types of viral hepatitis are hepatitis D and E and are less frequently encountered Cirrhosis results from chronic liver disease, and is characterized by advanced fibrosis, scarring, and formation of regenerative nodules leading to architectural distortion.In the past cirrhosis was generally thought to be irreversible but recent studies have shown that treatments aimed at the underlying cause especially in earlier stages of the disease can improve or even reverse fibrosis Since its discovery, hepatitis C virus (HCV) has been a constant burden for global health, with 3 to 4 million new infections each year and an overall number of 130-170 million infected people in the world New direct acting antiviral regimens (DAA) have changed the landscape of treatment of chronic hepatitis C DAA provide important advantages, including higher efficacy, shorter duration of treatment and an optimal safety profile Place of the study in patient admitted to Tropical Medicine and Gastroenterology Department, Sohag University Hospital Type of the study The study will be conducted in two stages The first one is a retrospective collection of the data from patients records during the period from Feburary 2017 to January 2018 and the second stage will include agroup of patients that will be admitted to Tropical Medicine and Gastroenterology Department within 6months after protocol acceptance Study period duration of study will be 6months after protocol acceptance Inclusion criteria:

Patients diagnosed with liver diseases(acute hepatitis, chronic hepatitis, liver cirrhosis, HCC and others) depending on clinical evidence of stigmata of liver disease (e.g. jaundice ,ascites ,palmar erythema , spider navi , etc),laboratory data and ultra sonographic features Methods Complete History Taking Clinical ExaminationLaboratory Investigations Abdominal Ultrasonography

DETAILED DESCRIPTION:
Liver disease accounts for approximately 2 million deaths per year worldwide, 1 million due to complications of cirrhosis and 1 million due to viral hepatitis and hepatocellular carcinoma Hepatitis is defined as inflammation of the liver that can result from a variety of causes such as heavy alcohol use, autoimmune, drugs, or toxins In the United States, the most common types of viral hepatitis are Hepatitis A, Hepatitis B, and Hepatitis C The other types of viral hepatitis are hepatitis D and E and are less frequently encountered Cirrhosis results from chronic liver disease, and is characterized by advanced fibrosis, scarring, and formation of regenerative nodules leading to architectural distortion.In the past cirrhosis was generally thought to be irreversible but recent studies have shown that treatments aimed at the underlying cause especially in earlier stages of the disease can improve or even reverse fibrosis Since its discovery, hepatitis C virus (HCV) has been a constant burden for global health, with 3 to 4 million new infections each year and an overall number of 130-170 million infected people in the world New direct acting antiviral regimens (DAA) have changed the landscape of treatment of chronic hepatitis C DAA provide important advantages, including higher efficacy, shorter duration of treatment and an optimal safety profile Place of the study in patient admitted to Tropical Medicine and Gastroenterology Department, Sohag University Hospital Type of the study The study will be conducted in two stages The first one is a retrospective collection of the data from patients records during the period from Feburary 2017 to January 2018 and the second stage will include agroup of patients that will be admitted to Tropical Medicine and Gastroenterology Department within 6months after protocol acceptance Study period duration of study will be 6months after protocol acceptance Inclusion criteria:

Patients diagnosed with liver diseases(acute hepatitis, chronic hepatitis, liver cirrhosis, HCC and others) depending on clinical evidence of stigmata of liver disease,laboratory data and ultra sonographic features Methods Complete History Taking Clinical ExaminationLaboratory Investigations Abdominal Ultrasonography

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with liver diseases depending on clinical evidence of stigmata of liver disease laboratory data and ultra sonographic features

Exclusion Criteria:

* Any patient without liver disease

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This study will include all patients admitted at Tropical Medicine and Gastroenterology Department, Sohag University Hospital diagnosed with liver diseases
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2022-09-15 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The different patterns of liver disease in patients admitted to Sohag University Hospital after the era of direct acting antiviral drugs | from 15 March 2022 to 15 September 2022

CONTACTS AND LOCATIONS:
Overall Officials: momena H Ahmed, master, Principal Investigator — Sohag University; Mona M Abdelrahman, MD, Study Director — Sohag University; Asmaa N Mohammed, MD, Study Chair — Sohag University

IPD SHARING:
Plan to Share IPD: No